CLINICAL TRIAL: NCT06457737
Title: The Performance of Posterior Partial Coverage Coronal Restorations Cemented Using Two Different Luting Systems. A Comparative Clinical Trial.
Brief Title: The Performance of Posterior Partial Coverage Coronal Restorations Luted With Two Differrent Systems.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20240137
Record Dates: First submitted 2024-06-03; First posted 2024-06-13 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Unsatisfactory or Defective Restoration of Tooth
Keywords: Endodontically treated teeth; Partial coverage; Ceramic restorations; Luting systems; Preheated composite; Dual cure adhesive resin cement
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Intervention Model Description: Split mouth study design, patients will be assigned to two different treatment protocols.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients who participated in the study and the assessor of the treatment outcome do not know the type of treatment procedure received.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preheated resin composite (IPS Empress Direct) group (Experimental): Endodontically treated teeth will be prepared to receive partial coverage ceramic restorations that will be luted with preheated composite.
  Interventions: Device: IPS Empress Direct
- Dual-cure adhesive resin cement (Bisco Duo-Link Universal) group (Experimental): Endodontically treated teeth will be prepared to receive partial coverage ceramic restorations that will be luted with dual-cure adhesive resin cement.
  Interventions: Device: Bisco Duo-Link Universal

INTERVENTIONS:
Device: IPS Empress Direct — Resin composite will be heated and used to lute a ceramic partial coverage restoration.
  Other Names: Ivoclar Vivadent, Schaan, Liechtenstein
  Arms: Preheated resin composite (IPS Empress Direct) group
Device: Bisco Duo-Link Universal — Dual cure adhesive resin cement will be used to lute a ceramic partial coverage restoration.
  Other Names: Bisco, USA
  Arms: Dual-cure adhesive resin cement (Bisco Duo-Link Universal) group

SUMMARY:
This study explores an alternative approach using a pre-heated restorative resin composite as a luting material of partial coverage restorations on upper and lower posterior teeth. It will follow a split-mouth design with 60 participants selected based on strict criteria. Assessment at 6 months and 1 year post-delivery utilizes a modified model of USPHS criteria, evaluating retention, color match, marginal discoloration, secondary caries, anatomical form, marginal adaptation, and surface roughness.

The null hypothesis:

The use of preheated resin composite for cementing partial coverage restoration will not result in significantly superior clinical performance when compared to that after using dual-cure resin cement.

DETAILED DESCRIPTION:
The adhesive cementation of ceramic partial coverage restorations is a technique-sensitive process essential for achieving optimal retention and marginal integrity. While dental resin cements are commonly used for adhesive luting of indirect ceramic restorations, concerns exist regarding their long-term reliability due to susceptibility to degradation over time and polymerization shrinkage-related issues.

This study explores an alternative approach using a pre-heated restorative resin composite as a luting material of partial coverage restorations on upper and lower posterior teeth, aiming to address these drawbacks. It will follow a split-mouth design with 60 participants selected based on strict criteria. The preparation and delivery appointments follow specific guidelines, incorporating the Morphology Driven Preparation Technique (MDPT). Assessment at 6 months and 1 year post-delivery utilizes a modified model of USPHS criteria, evaluating retention, color match, marginal discoloration, secondary caries, anatomical form, marginal adaptation, and surface roughness.

The objectives of this clinical trial are to evaluate the clinical performance of posterior partial coverage coronal restorations utilizing two different luting systems (preheated resin-based composite versus conventional dual-cure resin cement) in a split-mouth study design.

ELIGIBILITY:
Inclusion Criteria:

* Consenting participants.
* Individuals aged 18 years and above with no systemic diseases that will affect their participation.
* Teeth of healthy periodontium.
* Teeth to be restored in normal occlusion with natural antagonist and adjacent teeth.
* Acceptable oral hygiene characterized by no gingivitis, calculus deposit or active carious lesions.
* Non-vital teeth will be included

Exclusion Criteria:

* Heavy occlusal contacts or signs of bruxism.
* Profound, chronic periodontitis
* Poor oral hygiene.
* Sustained dentin hypersensitivity.
* Systemic disease or severe medical complications or taking anti-inflammatory, analgesic, or psychotropic drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation of the performance of restoration adaptation of posterior partial coverage ceramic restoration. | 1 year
  Clinical examination and evaluation of the adaptation quality of partial coverage restorations according to the United States Public Health Service (USPHS) criteria as Alpha, Beta, Charlie, Delta and Echo.
  Alpha score means: restoration contour is continuous with the existing anatomical margin of the tooth.
  Beta score means: restoration is slightly under or over contoured.
  Charlie score means: marginal overhang or tooth structure (dentin or enamel) is exposed.
  Delta score means: restoration is missing, or traumatic occlusion, or restoration causes pain.
Clinical evaluation of the presence or absence of caries adjacent to posterior partial coverage ceramic restoration. | 1 year
  Clinical examination and evaluation of the caries presence of partial coverage restorations according to the United States Public Health Service (USPHS) criteria as Alpha, Beta.
  Alpha score means: No visible caries
  Beta score means: caries present
Clinical evaluation of the performance of marginal adaptation of posterior partial coverage ceramic restoration. | 1 year
  Clinical examination and evaluation of the marginal adaptation quality of partial coverage restorations according to the United States Public Health Service (USPHS) criteria as Alpha, Beta, Charlie, Delta.
  Alpha score means: Excellent continuity at resin-enamel interface, no ledge formation, no discoloration
  Beta score means: Slight discoloration at resin-enamel interface; ledge at interafce.
  Charlie score means: Moderate discoloration at resin-enamel interface measuring 1mm or greater.
  Delta score means: Recurrent caries at margins.
Clinical evaluation of surface staining of posterior partial coverage ceramic restoration. | 1 year
  Clinical examination and evaluation of the presence or absence of surface staining of partial coverage restorations according to the United States Public Health Service (USPHS) criteria as Alpha, Beta.
  Alpha score means: staining absent
  Beta score means: staining present
Clinical evaluation of contact points of posterior partial coverage ceramic restoration. | 1 year
  Clinical examination and evaluation of the contact points quality of partial coverage restorations according to the United States Public Health Service (USPHS) criteria as Alpha, Beta.
  Alpha score means: contact point present
  Beta score means: contact point absent.
Clinical evaluation of fracture of posterior partial coverage ceramic restoration. | 1 year
  Clinical examination and evaluation of the structural integrity endurance of partial coverage restorations according to the United States Public Health Service (USPHS) criteria as Alpha, Beta, Charlie, Delta, Echo.
  Alpha score means: No fracture of the restoration.
  Beta score means: Small chipping (1/4 of restoration)
  Charlie score means: Moderate chipping (1/2 of restoration)
  Delta score means: Severe chipping (3/4 of restoration)
  Echo score means: loss of the restoration.
Clinical evaluation of wear of posterior partial coverage ceramic restoration. | 1 year
  Clinical examination and evaluation of the wear presence or absence of partial coverage restorations according to the United States Public Health Service (USPHS) criteria as Alpha, Beta.
  Alpha score means: absence of wear.
  Beta score means: wear present.
Radiographic evaluation of the performance of restoration adaptation of posterior partial coverage ceramic restoration. | 1 year
  Radiographic examination and evaluation of the adaptation quality of partial coverage restorations according to the United States Public Health Service (USPHS) criteria as Alpha, Beta, Charlie, Delta and Echo.
  Alpha score means: restoration contour is continuous with the existing anatomical margin of the tooth.
  Beta score means: restoration is slightly under or over contoured.
  Charlie score means: marginal overhang or tooth structure (dentin or enamel) is exposed.
  Delta score means: restoration is missing.
Radiographic evaluation of the presence or absence of caries adjacent to posterior partial coverage ceramic restoration. | 1 year
  Radiographic examination and evaluation of the caries presence of partial coverage restorations according to the United States Public Health Service (USPHS) criteria as Alpha, Beta.
  Alpha score means: No visible caries
  Beta score means: caries present
Radiographic evaluation of marginal adaptation of posterior partial coverage ceramic restoration. | 1 year
  Radiographic examination and evaluation of the marginal adaptation quality of partial coverage restorations according to the United States Public Health Service (USPHS) criteria as Alpha, Beta, Charlie, Delta.
  Alpha score means: Excellent continuity at resin-enamel interface, no ledge formation, no discoloration
  Beta score means: Slight discoloration at resin-enamel interface; ledge at interafce.
  Charlie score means: Moderate discoloration at resin-enamel interface measuring 1mm or greater.
  Delta score means: Recurrent caries at margins.

CONTACTS AND LOCATIONS:
Overall Officials: Zakereyya SM Albashaireh, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No
A consent has to be obtained from the faculty of graduate studies for sharing data as data form part of graduate students thesis.

REFERENCES:
- [Background] Veneziani M. Posterior indirect adhesive restorations: updated indications and the Morphology Driven Preparation Technique. Int J Esthet Dent. 2017;12(2):204-230. PMID 28653051
- [Background] Rickman LJ, Padipatvuthikul P, Chee B. Clinical applications of preheated hybrid resin composite. Br Dent J. 2011 Jul 22;211(2):63-7. doi: 10.1038/sj.bdj.2011.571. PMID 21779058
- [Background] Ayub KV, Santos GC Jr, Rizkalla AS, Bohay R, Pegoraro LF, Rubo JH, Santos MJ. Effect of preheating on microhardness and viscosity of 4 resin composites. J Can Dent Assoc. 2014;80:e12. PMID 24598328
- [Background] Mundim FM, Garcia Lda F, Cruvinel DR, Lima FA, Bachmann L, Pires-de-Souza Fde C. Color stability, opacity and degree of conversion of pre-heated composites. J Dent. 2011 Jul;39 Suppl 1:e25-9. doi: 10.1016/j.jdent.2010.12.001. Epub 2010 Dec 14. PMID 21163324
- [Background] da Costa JB, Hilton TJ, Swift EJ Jr. Critical appraisal: preheating composites. J Esthet Restor Dent. 2011 Aug;23(4):269-75. doi: 10.1111/j.1708-8240.2011.00461.x. Epub 2011 Jun 22. PMID 21806761
- [Background] Marcondes RL, Lima VP, Barbon FJ, Isolan CP, Carvalho MA, Salvador MV, Lima AF, Moraes RR. Viscosity and thermal kinetics of 10 preheated restorative resin composites and effect of ultrasound energy on film thickness. Dent Mater. 2020 Oct;36(10):1356-1364. doi: 10.1016/j.dental.2020.08.004. Epub 2020 Sep 1. PMID 32888725
- [Background] Patussi AFC, Ramacciato JC, da Silva JGR, Nascimento VRP, Campos DES, de Araujo Ferreira Munizz I, de Souza GM, Lima RBW. Preheating of dental composite resins: A scoping review. J Esthet Restor Dent. 2023 Jun;35(4):646-656. doi: 10.1111/jerd.12991. Epub 2022 Dec 7. PMID 36478368
- [Background] Magne P, Razaghy M, Carvalho MA, Soares LM. Luting of inlays, onlays, and overlays with preheated restorative composite resin does not prevent seating accuracy. Int J Esthet Dent. 2018;13(3):318-332. PMID 30073216
- [Background] Coelho NF, Barbon FJ, Machado RG, Boscato N, Moraes RR. Response of composite resins to preheating and the resulting strengthening of luted feldspar ceramic. Dent Mater. 2019 Oct;35(10):1430-1438. doi: 10.1016/j.dental.2019.07.021. Epub 2019 Aug 3. PMID 31387743
- [Background] Gresnigt MMM, Ozcan M, Carvalho M, Lazari P, Cune MS, Razavi P, Magne P. Effect of luting agent on the load to failure and accelerated-fatigue resistance of lithium disilicate laminate veneers. Dent Mater. 2017 Dec;33(12):1392-1401. doi: 10.1016/j.dental.2017.09.010. Epub 2017 Nov 1. PMID 29079354
- [Background] Skapska A, Komorek Z, Cierech M, Mierzwinska-Nastalska E. Comparison of Mechanical Properties of a Self-Adhesive Composite Cement and a Heated Composite Material. Polymers (Basel). 2022 Jun 30;14(13):2686. doi: 10.3390/polym14132686. PMID 35808732
- [Background] Falacho RI, Marques JA, Palma PJ, Roseiro L, Caramelo F, Ramos JC, Guerra F, Blatz MB. Luting indirect restorations with resin cements versus composite resins: Effects of preheating and ultrasound energy on film thickness. J Esthet Restor Dent. 2022 Jun;34(4):641-649. doi: 10.1111/jerd.12851. Epub 2021 Dec 13. PMID 34897958
- [Background] Goujat A, Abouelleil H, Colon P, Jeannin C, Pradelle N, Seux D, Grosgogeat B. Marginal and internal fit of CAD-CAM inlay/onlay restorations: A systematic review of in vitro studies. J Prosthet Dent. 2019 Apr;121(4):590-597.e3. doi: 10.1016/j.prosdent.2018.06.006. Epub 2018 Dec 1. PMID 30509548
- [Background] Schmidlin PR, Zehnder M, Schlup-Mityko C, Gohring TN. Interface evaluation after manual and ultrasonic insertion of standardized class I inlays using composite resin materials of different viscosity. Acta Odontol Scand. 2005 Aug;63(4):205-12. doi: 10.1080/00016350510019973. PMID 16040442
- [Background] Magne P. Immediate dentin sealing: a fundamental procedure for indirect bonded restorations. J Esthet Restor Dent. 2005;17(3):144-54; discussion 155. doi: 10.1111/j.1708-8240.2005.tb00103.x. PMID 15996383
- See also: ISO-4049:2019 standard: The polymer-based luting materials covered by this document are intended for use in the cementation or fixation of restorations and appliances such as inlays, onlays, veneers, crowns and bridges. — https://www.iso.org/standard/67596.html
- See also: Sealed Envelope Ltd. 2012. Power calculator for binary outcome superiority trial. [Online] — https://www.sealedenvelope.com/power/binary-superiority